CLINICAL TRIAL: NCT04210999
Title: Is Supervised or Homebased Resistance Training the Best Treatment for Chronic Achilles Tendinopathy? And When Needed is Supplement Treatment With Either Corticosteroid or High Volume Injection the Best Choice
Brief Title: Resistance Training and Injection Treatment for Chronic Achilles Tendinopathy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Simon Doessing, M.D., PhD, Senior Surgeon, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-19040270
Record Dates: First submitted 2019-12-22; First posted 2019-12-26 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Achilles Tendinopathy

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Homebased resistance training (Experimental): Resistance training at home instructed via a smart phone training app and avoidance of pain aggravating activities for 3 months
  Interventions: Other: Homebased resistance training
- Supervised resistance training (Active Comparator): Heavy slow resistance training in the gym instructed by a physiotherapist and avoidance of pain aggravating activities for 3 months
  Interventions: Other: Supervised heavy slow resistance training

INTERVENTIONS:
Other: Homebased resistance training — Resistance training at home instructed via a smart phone training app
  Arms: Homebased resistance training
Other: Supervised heavy slow resistance training — Heavy slow resistance training in the gym instructed by a physiotherapist
  Arms: Supervised resistance training

SUMMARY:
Achilles tendinopathy is a common and often long-lasting injury among exercising individuals.

The primary purpose of the study is to compare treatment with supervised or homebased resistance training. The secondary purpose is to compare treatment with either corticosteroid or High Volume Injection (HVI) for those patients not responding to the primary treatment.

The tertiary purpose is to evaluate the effect of surgery in those patients not responding to the primary and the secondary treatment.

It is hypothesized that:

1. Homebased resistance training is as effective as supervised resistance training for treating chronic achilles tendinopathy
2. HVI injection is better than CS injection for those patients not responding sufficiently to treatment 1
3. Surgery improves symptoms in patients not responding to treatment 1 and treatment 2

Study 1: 90 patients between 18 and 65 years of age with achilles tendinopathy for at least 3 months are randomly assigned to either A. Resistance training at home instructed via a smart phone training app and avoidance of pain aggravating activities for 3 months B. Heavy slow resistance training in the gym instructed by a physiotherapist and avoidance of pain aggravating activities for 3 months

Outcomes are change in patient reported outcome (VISA-A) from baseline to 3 and 6 months, ultrasound measured thickness and dopler activity of the achilles tendon, self reported activity level in percentage of the pre injury activity level.

After the 3-month training intervention, and for the following 9 months, those patients that not are satisfied with the outcome will have the opportunity to participate in the second part of the study.

Study 2: Patients from study 1 which not are satisfied with the outcome are randomly assigned to either

A. Same training intervention continued + High Volume Injection (HVI) B. Same training intervention continued + corticosteroid injection

After the 4-month and for the following 8 months, those patients that not are satisfied with the outcome will have the opportunity to participate in the third part of the study.

Study 3: Patients from study 2 which not are satisfied with the outcome are operated

DETAILED DESCRIPTION:
Achilles tendinopathy is a common and often long-lasting injury among exercising individuals. Treatment options typically include rest from high load weight bearing activities, resistance training, injections with corticosteroid (CS) or High Volume Injection (HVI) and surgery.

The primary purpose of the study is to compare treatment with supervised or homebased resistance training.

The secondary purpose is to compare treatment with either corticosteroid or High Volume Injection (HVI) for those patients not responding to the primary treatment.

The tertiary purpose is to evaluate the effect of surgery in those patients not responding to the primary and the secondary treatment.

It is hypothesized that:

4. Homebased resistance training is as effective as supervised resistance training for treating chronic achilles tendinopathy (RCT, non-inferiority design).

5. HVI injection is better than CS injection for those patients not responding sufficiently to treatment 1. (RCT, superiority design).

6. Surgery improves symptoms in patients not responding to treatment 1. and treatment 2. (prospective cohort).

Study 1: 90 patients with achilles tendinopathy are randomly assigned to either

C. Resistance training at home instructed via a smart phone training app and avoidance of pain aggravating activities for 3 months D. Heavy slow resistance training in the gym instructed by a physiotherapist and avoidance of pain aggravating activities for 3 months

Inclusion criteria

* Pain from the achilles tendon either unilateral or bilateral for at least 3 months
* Achilles tendinopathy in the tendon midsubstance verified by ultrasound
* Between 18 and 65 years of age
* For patients with unilaterale symptoms the symptomatic tendon must be at least 20% thicker than on the asymptomatic side or more than 7 mm thick
* For patients with bilateral symptoms the achilles tendons must have diameters above 7 mm Exclusion criteria
* Prior surgery in the leg with the exception of knee arthroscopy
* Known medial conditions including diabetes or rheumatologic diseases
* Taking pain medication regularly
* Injection therapy for treatment of achilles tendinopathy within the last 6 months

Patients are stratified based on the severity of symptoms (below or above 50 on VISA-A) and duration of symptoms (shorter or longer than 1 year)

ELIGIBILITY:
Inclusion Criteria:

* Pain from the achilles tendon either unilateral or bilateral for at least 3 months
* Achilles tendinopathy in the tendon midtsubstance verified by ultrasound
* Between 18 and 65 years of age
* For patients with unilaterale symptoms the symptomatic tendon must be at least 20% thicker than on the asymptomatic side or more than 7 mm thick
* For patients with bilateral symptoms the achilles tendons must have diameters above 7 mm

Exclusion Criteria:

* Prior surgery in the leg with the exception of knee artroscopy
* Known medial conditions including diabetes or rheumatologic diseases
* Taking pain medication regularly
* Injection therapy for treatment of achilles tendinopati within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-04-05 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in The Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A). | After 3 and 6 months in study 1. After 6 months in study 2. After 6 and 12 months in study 3.
  VISA-A is a patient reported outcome measure (PROM). Change from baseline is measured and reported. The scale ranges from 0-100 points. Higher score meaning a better outcome.

SECONDARY OUTCOMES:
Evaluation of treatment effect measured on an 11-point Likert scale. | After 1, 2, 3, 6, 9 and 12 months in study 1 and study 2. After 3, 6 and 12 months in study 3.
  The Likert scale used is an 11-point scale ranging from -5 to +5. +5 is cured and -5 is much worsened, 0 is the status when entering the study.
Change from baseline in The Victorian Institute of Sports Assessment - Achilles Questionnaire (VISA-A). | After 1, 2, 9 and 12 months in study 1. After 1, 3, 6, 9 and 12 months in study 2. After 3 months in study 3.
  VISA-A is a patient reported outcome measure (PROM). Change from baseline is measured and reported. The scale ranges from 0-100 points. Higher score meaning a better outcome.
Evaluation of the training experience measured on a Likert scale. | After 3 months in study 1. After 3 months in study 2.
  The Likert scale used is an 11-point scale ranging from -5 to +5. +5 is very inspiring/motivating, -5 is very uninspiring/boring, 0 representing the status when entering the study.
Ultrasonographic measurement of achilles tendon thickness and doppler activity. | After 0, 1, 2, 3, 6 and 12 months in study 1 and study 2. After 3, 6 and 12 months in study 3.
  Ultrasonographic measurement of achilles tendon thickness and doppler activity is measured relative to the baseline values.
Patient self reported activity level in percentage of the pre-injury activity level. | After 6, 9 and 12 months in study 1 and study 2. After 3, 6 and 12 months in study 3.
  Self reported activity level in percentage of the pre-injury activity level is reported.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjaer, MD. PhD, Study Director — University of Copenhagen and Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-11-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT04210999/SAP_000.pdf